CLINICAL TRIAL: NCT00271375
Title: Evaluating the Carter Institute Caregiver Education Program at the VA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: E4044-R; IRB 2005-050240 (Other: Atlanta VAMC); IRB 278-2005 (Other: Emory University IRB)
Record Dates: First submitted 2005-12-29; First posted 2005-12-30 (Estimated); Results first posted 2016-05-30 (Estimated); Last update posted 2016-05-30 (Estimated); Status verified 2016-04

CONDITIONS: Caregivers
Keywords: Age; Caregivers; Family; Intervention Studies

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1: Caring for you, Caring for me Educational Intervention (Experimental): Educational Intervention
  Interventions: Behavioral: Caring For You, Caring For Me
- Arm 2: Caring for you, caring for me + social worker (Experimental): Educational + Social Work Intervention
  Interventions: Behavioral: Caring for you, caring for me + social worker
- Arm 3: Control group usual care (Placebo Comparator): Control group usual care
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Caring For You, Caring For Me — 5-week Education and Support Program for Caregivers of older adults.
  Arms: Arm 1: Caring for you, Caring for me Educational Intervention
Behavioral: Caring for you, caring for me + social worker — 5-week Education and Support Program for Caregivers of older adults.+ augmentation with social worker
  Arms: Arm 2: Caring for you, caring for me + social worker
Behavioral: Control — Control group usual care
  Arms: Arm 3: Control group usual care

SUMMARY:
This project implemented and evaluated the Rosalyn Carter Institute's (RCI's) educational and support program for caregivers, "Caring for You, Caring for Me." Specifically, it examined effects of the program upon family caregivers to older adults in the Atlanta area and elderly Veterans receiving outpatient primary care at the Atlanta Veterans Affairs Medical Center (VAMC).

DETAILED DESCRIPTION:
Primary objectives of the research were:

1. to evaluate user satisfaction with and perceived utility of the "Caring for You, Caring for Me" caregiver educational program among formal (VHA staff) and informal (family) caregivers who undergo the program;
2. to assess effects of the program upon psychosocial and physical well-being of informal caregivers over a 1-year period .

ELIGIBILITY:
Inclusion Criteria:

* Family members of Veterans aged 65+ years and receiving care through the Atlanta VAMC's Clinic and Atlanta area.
* Must be the primary caregiver to someone 55 and over.
* Must have been assisting with at least one activity of daily living (ADL) for at least 6 months prior to beginning the intervention.

Exclusion Criteria:

* Caregivers are automatically excluded if veteran has a terminal illness with six months or less to live.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2005-10; Primary Completion 2009-08 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Griffiths, PhD, Principal Investigator — Atlanta VAMC
Locations (1):
- VA Medical Center, Decatur, Decatur, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Caring for You, Caring for me Educational Intervention: Caring For You, Caring For Me: 5-week Education and Support Program for Caregivers of older adults.
- Caring for You, Caring for me + Social Worker (Educational Int: Caring for you, caring for me + social worker: 5-week Education and Support Program for Caregivers of older adults.+ augmentation with social worker
- Control Group Usual Care: Control: Control group usual care
Period: Overall Study
Arm/Group | Caring for You, Caring for me Educational Intervention | Caring for You, Caring for me + Social Worker (Educational Int | Control Group Usual Care
Started | 114 | 83 | 57
Completed | 114 | 83 | 57
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Caring for You, Caring for me Educational Intervention | Caring for You, Caring for me + Social Worker (Educational Int | Control Group Usual Care | Total
Number analyzed (Participants) | 114 | 83 | 57 | 254
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age
  Years | 66.9 (11.0) | 63.4 (11.7) | 61.1 (9.8) | 64.69 (11.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111 | 76 | 51 | 238
  Male | 3 | 7 | 6 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 38 | 31 | 24 | 93
  White | 74 | 52 | 30 | 156
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate User Satisfaction With and Perceived Utility of the "Caring for You, Caring for Me" Caregiver Educational Program Among Formal (VHA Staff) and Informal (Family) Caregivers Who Undergo the Program
Description: This question addresses user satisfaction, in terms of caregiving perceived utility of the education program, as well as their actual use of knowledge and skills gained in their caregiving situation.
Time Frame: 18 Months
Population: User evaluation of the "Caring for you, Caring for me" education program. Data for participants in the "Caring for you, Caring for me" education program only and "Caring for you, Caring for me" education program+ Social Work were combined during data collection. Only 71 participants provided results. No data was collected from control group.
Measure: Number; unit: participants
Groups:
- Overall Evaluation: Caring For You, Caring For Me: 5-week Education and Support Program for Caregivers of older adults.
Arm/Group | Overall Evaluation
Number analyzed (Participants) | 71
participants
  Excellent | 31
  Very Good | 32
  Good | 8
  Fair | 0
  Poor | 0

2. Secondary Outcome: Subjective Health
Description: Subjective Health was assessed using one of the eight subscales from the Medical Outcomes Study Health Survey Short Form (SF-36) which looked at the how the respondent (caregiver) perceived their own health currently and compared to a year ago. Two items were based on a 5-point Likert scale (1 =Excellent and 5= Poor) with a total scale range between 1 and 5. Mean scores were calculated by finding the total sum divided by the total number of items, with higher scores indicating poorer outcomes. Calculations were completed at each time interval (baseline, 6month follow-up, and 12month follow-up) and for each study arm (Arm 1, Arm 2 and Arm 3).
Time Frame: Baseline, 6 Month Follow-up, 12 Month Follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Arm 2: Caring for You, Caring for me + Social Worker (Educati: Caring for you, caring for me + social worker: 5-week Education and Support Program for Caregivers of older adults.+ augmentation with social worker
Arm/Group | Arm 1: Caring for You, Caring for me Educational Intervention | Arm 2: Caring for You, Caring for me + Social Worker (Educati | Arm 3: Control Group Usual Care
Number analyzed (Participants) | 114 | 83 | 57
units on a scale
  Baseline | 3.49 (.83) | 3.68 (.77) | 3.37 (.64)
  6 Month Follow-up | 3.11 (.62) | 3.17 (.58) | 3.12 (.59)
  12 month Follow-up | 3.06 (.67) | 3.19 (.72) | 3.05 (.44)

3. Secondary Outcome: Physical Role Function
Description: Physical Role Function was assessed using one of the eight subscales from the Medical Outcomes Study Health Survey Short Form (SF-36) which looked at how emotional or physical issues interfered with everyday social roles of the caregiver. 4 items were scored on a 5-point Likert scale (1 = All of the time and 5= None of the time) with total scale range between 1 and 5. Mean scores were calculated by finding the total sum divided by the total item number, with lower scores indicating poorer outcome. Calculations were completed at each time interval (baseline, 6month follow-up, and 12month follow-up) and for each study arm (Arm 1, Arm 2 and Arm 3).
Time Frame: Baseline, 6 Month Follow-up, 12 Month Follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: Caring for You, Caring for me Educational Intervention | Arm 2: Caring for You, Caring for me + Social Worker (Educati | Arm 3: Control Group Usual Care
Number analyzed (Participants) | 114 | 83 | 57
units on a scale
  Baseline | 3.88 (1.06) | 4.33 (1.01) | 3.90 (0.93)
  6 Month Follow-up | 3.90 (.98) | 4.11 (0.94) | 4.16 (0.88)
  12 Month Follow-up | 3.80 (0.98) | 4.20 (0.98) | 4.19 (0.77)

4. Secondary Outcome: Physical Function
Description: Physical function was assessed using one of the eight subscales from the Medical Outcomes Study Health Survey Short Form (SF-36) which is represented by 10 items tapping basic functional abilities of the caregiver (Does their health limit them in the following activities). 10 items were scored on a 3-Point Likert Scale with 1= Limited A lot and 3= Not Limited and total scale range between 1 and 3. Mean scores were calculated by finding the total sum divided by the total item number, with lower scores indicating poorer outcome. Calculations were completed at each time interval (baseline, 6month follow-up, and 12month follow-up) and for each study arm (Arm 1, Arm 2 and Arm 3).
Time Frame: Baseline, 6 Month Follow-up, 12 Month Follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: Caring for You, Caring for me Educational Intervention | Arm 2: Caring for You, Caring for me + Social Worker (Educati | Arm 3: Control Group Usual Care
Number analyzed (Participants) | 114 | 83 | 57
units on a scale
  Baseline | 2.36 (.52) | 2.52 (.48) | 2.58 (.40)
  6 Month Follow-up | 2.39 (.51) | 2.64 (.41) | 2.68 (.37)
  12 Month Follow-up | 2.31 (.57) | 2.62 (.45) | 1.57 (.38)

5. Secondary Outcome: Depressive Symptoms
Description: Depression symptoms were assessed using the Center for Epidemiological Studies Depression Scale (CES-D Short Form). The CES-D is a 10 Question Scale with total scores ranging from 0-30. Mean scores were calculated by finding the total sum divided by the total number of participants. Any score equal to or above 10 is considered depressed. Calculations were completed at each time interval (baseline, 6month follow-up, and 12month follow-up) and for each study arm (Arm 1, Arm 2 and Arm 3).
Time Frame: Baseline, 6 Month Follow-up, 12 Month Follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: Caring for You, Caring for me Educational Intervention | Arm 2: Caring for You, Caring for me + Social Worker (Educati | Arm 3: Control Group Usual Care
Number analyzed (Participants) | 114 | 83 | 57
units on a scale
  Baseline | 10.54 (9.67) | 9.96 (7.97) | 12.18 (12.64)
  6 Month Follow-up | 9.27 (7.96) | 8.29 (8.07) | 12.47 (11.79)
  12 Month Follow-up | 11.37 (9.37) | 7.50 (7.18) | 11.41 (9.42)

6. Secondary Outcome: Caregiver Burden
Description: Caregiver Burden was assessed using one of the five subscales from the revised Caregiver Appraisal Scale (CAS) through 9-items based on a 5-point likert scale with (1 = Never and 5= Nearly always). Mean for the total scores, calculated as the total sum divided by the number of participants, where scores could range from 9 to 45 were calculated, with higher scores indicating poorer outcomes. Calculations were completed at each time interval (baseline, 6month follow-up, and 12month follow-up) and for each study arm (Arm 1, Arm 2 and Arm 3).
Time Frame: Baseline, 6 Month Follow-up, 12 Month Follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: Caring for You, Caring for me Educational Intervention | Arm 2: Caring for You, Caring for me + Social Worker (Educati | Arm 3: Control Group Usual Care
Number analyzed (Participants) | 114 | 83 | 57
units on a scale
  Baseline | 23.02 (8.62) | 23.93 (8.27) | 23.41 (8.48)
  6 Month Follow-up | 22.61 (6.61) | 22.07 (7.43) | 22.65 (8.29)
  12 Month Follow-up | 23.68 (8.44) | 21.57 (7.69) | 21.06 (8.18)

7. Secondary Outcome: Caregiver Satisfaction
Description: Caregiver Satisfaction was assessed using one of the five subscales from the revised Caregiver Appraisal Scale (CAS) through 6-items based on a 5-point likert scale with (1 = Disagree A lot and 5= Agree A lot). Mean for the total scores, calculated as the total sum divided by the number of participants, where scores could range from 6 to 30 were calculated, with higher scores indicating poorer outcomes. Calculations were completed at each time interval (baseline, 6month follow-up, and 12month follow-up) and for each study arm (Arm 1, Arm 2 and Arm 3).
Time Frame: Baseline, 6 Month Follow-up, 12 Month Follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: Caring for You, Caring for me Educational Intervention | Arm 2: Caring for You, Caring for me + Social Worker (Educati | Arm 3: Control Group Usual Care
Number analyzed (Participants) | 114 | 83 | 57
units on a scale
  Baseline | 23.15 (4.26) | 23.5 (5.44) | 26.00 (3.16)
  6 Month Follow-up | 23.02 (4.64) | 23.43 (4.98) | 25.88 (3.81)
  12 Month Follow-up | 22.83 (4.97) | 23.50 (4.81) | 25.18 (4.63)

8. Secondary Outcome: Caregiver Mastery
Description: Caregiver Mastery was assessed using one of the five subscales from the revised Caregiver Appraisal Scale (CAS) through a 4-item question assessing a sense of doing a good job of care provision based on a 5-point likert scale with (5= Agree A lot and 1= Disagree A lot). Mean for the total scores, calculated as the total sum divided by the number of participants, where scores could range from 5 to 20 were calculated, with higher scores indicating poorer outcome. Calculations were completed at each time interval (baseline, 6month follow-up, and 12month follow-up) and for each study arm (Arm 1, Arm 2 and Arm 3).
Time Frame: Baseline, 6 Month Follow-up, 12 Month Follow-up
Measure: Median (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: Caring for You, Caring for me Educational Intervention | Arm 2: Caring for You, Caring for me + Social Worker (Educati | Arm 3: Control Group Usual Care
Number analyzed (Participants) | 114 | 83 | 57
units on a scale
  Baseline | 13.51 (3.50) | 13.25 (3.34) | 11.59 (3.06)
  6 Month Follow-up | 10.90 (2.41) | 11.21 (2.13) | 9.59 (1.73)
  12 Month Follow-up | 6.88 (2.23) | 7.04 (1.86) | 6.24 (2.28)

9. Secondary Outcome: Caregiver Efficacy
Description: Caregiver Efficacy was assessed using the RIS Eldercare Self Efficacy Scale (RIS) a 10-item inventory addressing family caregiver's perception of their own ability to manage care provision challenges in the areas of relationship with the care recipient, instrumental care provision, and self-soothing (managing the strains of care provision) based on a 5-point likert scale with (1 = Im certain I CANNOT Do This and 5= Im certain I CAN Do This) with a total score range between1 and 5. Mean scores were calculated by finding the total sum divided by the total item number, higher scores indicating better outcome. Calculations were completed at each time interval (baseline, 6month follow-up, and 12month follow-up) and for each study arm (Arm 1, Arm 2 and Arm 3).
Time Frame: Baseline, 6 Month Follow-up, 12 Month Follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: Caring for You, Caring for me Educational Intervention | Arm 2: Caring for You, Caring for me + Social Worker (Educati | Arm 3: Control Group Usual Care
Number analyzed (Participants) | 114 | 83 | 57
units on a scale
  Baseline | 4.15 (0.65) | 4.16 (0.52) | 4.78 (0.41)
  6 Month Follow-up | 4.15 (0.47) | 4.18 (0.52) | 4.15 (0.55)
  12 Month Follow-up | 4.09 (0.52) | 4.22 (0.50) | 4.17 (0.47)

10. Secondary Outcome: Personal Mastery
Description: Caregiver Personal Mastery was assessed using the Personal Mastery Scale which afforded a general measure of self-perceived ability to manage stressors and effect change in one's life through a 7-item question based on a 5-point likert scale with (5 = Agree A lot and 1= Disagree A lot) and a total score range between 1 and 5. Mean scores were calculated by finding the total sum divided by the total item number, with higher scores indicating poorer outcome. Calculations were completed at each time interval (baseline, 6month follow-up, and 12month follow-up) and for each study arm (Arm 1, Arm 2 and Arm 3).
Time Frame: Baseline, 6 Month Follow-up, 12 Month Follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: Caring for You, Caring for me Educational Intervention | Arm 2: Caring for You, Caring for me + Social Worker (Educati | Arm 3: Control Group Usual Care
Number analyzed (Participants) | 114 | 83 | 57
units on a scale
  Baseline | 3.60 (0.73) | 3.84 (0.65) | 3.50 (0.74)
  6 Month Follow-up | 3.64 (0.76) | 3.90 (0.77) | 3.56 (0.54)
  12 Month Follow-up | 3.70 (0.79) | 3.89 (0.76) | 3.52 (0.86)

11. Secondary Outcome: Perceived Social Support
Description: Caregiver Perceived Social Support was assessed using the Medical Outcomes Study Social Support Survey (MOS-SSS) a 19-item scale that taps perceived emotional/informational, tangible, and affectionate support, and positive social interaction based on a 5-point likert scale with (1 = None of the time and 5= All of the time) with total score range between 1 and 5. Mean scores were calculated by finding the total sum divided by the total item number, with higher scores indicating better outcome. Calculations were completed at each time interval (baseline, 6month follow-up, and 12month follow-up) and for each study arm (Arm 1, Arm 2 and Arm 3).
Time Frame: Baseline, 6 Month Follow-up, 12 Month Follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: Caring for You, Caring for me Educational Intervention | Arm 2: Caring for You, Caring for me + Social Worker (Educati | Arm 3: Control Group Usual Care
Number analyzed (Participants) | 114 | 83 | 57
units on a scale
  Baseline | 3.70 (0.81) | 3.77 (0.90) | 3.70 (0.76)
  6 Month Follow-up | 3.65 (0.76) | 3.81 (0.87) | 3.81 (0.92)
  12 Month Follow-up | 3.72 (0.81) | 3.79 (0.90) | 3.51 (0.77)

ADVERSE EVENTS:
Arm/Group | Arm 1: Caring for You, Caring for me Educational Intervention | Arm 2: Caring for You, Caring for me + Social Worker (Educati | Arm 3: Control Group Usual Care
Serious Adverse Events (participants affected / at risk) | 0/114 | 0/83 | 0/57
Other Adverse Events (participants affected / at risk) | 0/114 | 0/83 | 0/57

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes